CLINICAL TRIAL: NCT04047264
Title: Intraoperative Microdialysis During Neurosurgery for Central Nervous System Malignancies
Brief Title: Feasibility of Intraoperative Microdialysis During Neurosurgery for Central Nervous System Malignancies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-004694; NCI-2021-02742 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-004694 (Other: Mayo Clinic Institutional Review Board); R37CA276851 (NIH); R61NS122096 (NIH)
Record Dates: First submitted 2019-07-29; First posted 2019-08-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Glioma; Glioblastoma; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms | interventions — Microdialysis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Basic Science (microdialysis) (Experimental): Patients undergo microdialysis over 30 minutes during standard of care biopsy or resection.
  Interventions: Procedure: Microdialysis; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Microdialysis — Undergo microdialysis
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging (MRI); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; NMR Imaging; Nuclear Magnetic Resonance Imaging (NMRI); nuclear magnetic resonance imaging; sMRI; Structural MRI

SUMMARY:
This clinical trial evaluates the use of microdialysis catheters during surgery to collect biomarkers, and studies the feasibility of intraoperative microdialysis during neurosurgery for central nervous system malignancies. A biomarker is a measurable indicator of the severity or presence of disease state. Information collected in this study may help doctors to develop new strategies to better diagnose, monitor, and treat brain tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine biomarkers of in situ gliomas across a diverse patient cohort using intra-operative microdialysis to sample extracellular metabolites.

SECONDARY OBJECTIVE:

I. Evaluate the yield and specificity of microdialysate D-2HG as a candidate tumor biomarker to differentiate between IDH-mutated and IDH-wildtype gliomas.

II. Identify biomarkers of tumor-associated processes including brain edema, brain infiltration with non-enhancing tumor, and tumor-associated hypoxia or necrosis.

III. Determine the contribution of blood-brain barrier disruption to metabolite abundance within enhancing gliomas.

EXPLORATORY/CORRELATIVE OBJECTIVES:

I. Perform untargeted metabolomics of tumor microdialysate to elucidate extracellular biomarkers reflective of human central nervous system malignancy subtype, grade, and tumor region.

II. Banking of microdialysate specimens for future analyses.

OUTLINE:

Patients undergo microdialysis over 30 minutes during standard of care biopsy or resection.

After completion of study, patients are followed up for 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of the following, based on clinical and radiographic evidence:

  * Any glioma
  * Metastatic brain tumor of any primary origin
  * Epileptic focus requiring surgical resection
* Planned neurosurgical procedure for purposes of biopsy or resection of suspected or previously diagnosed brain tumor (primary or metastatic) or epileptic focus as part of routine clinical care
* Willing to undergo neurosurgical resection or biopsy at Mayo Clinic (Rochester, Minnesota [MN])
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Vulnerable populations: pregnant women, prisoners or the mentally handicapped
* Patients who are not appropriate candidates for surgery due to current or past medical history or uncontrolled concurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 42 days
  Will be assessed by evaluating the proportion of patients who: (2) develop persistent adverse events deemed related (possibly, probably, definitely) to the insertion or use of microdialysate catheters. Attribution of neurologic deficit will typically be considered unlikely unless there is evidence of intra-operative intracranial hemorrhage that the surgeon deems to be attributable to use of the microdialysis catheter. Adverse events will be measured by Common Terminology Criteria for Adverse Events 5.0.
Targeted metabolomics | Up to 42 days
  Metabolites within each region of tumor to brain-adjacent-to tumor within a patient compared. Metabolites from patients without central nervous system malignancies averaged across the epileptic foci group and descriptively compared to the areas from patients with gliomas.

SECONDARY OUTCOMES:
Microdialysate D-2HG | Up to 42 days
  Concentrations of D-2HG in microdialysate will be descriptively compared between patients with IDH mutated gliomas and those with IDH wildtype gliomas.
Non-enhancing (FLAIR)- region metabolites | Up to 42 days
  Metabolites of non-glioma, edema-associated FLAIR region of metastatic tumors descriptively compared to those within non-enhancing FLAIR gliomas.
Necrotic core metabolites | Up to 42 days
  The relative contribution of tumor cellularity versus blood-brain barrier disruption to metabolite production and loss determined by comparing metabolites within the necrotic tumor to those found within the enhancing tumor and brain -adjacent-to-tumor.

OTHER OUTCOMES:
Microdialysate oncometabolites | Up to 42 days
  Will be assessed by untargeted metabolomic analyses will be tabulated and evaluated for hypothesis generation.

CONTACTS AND LOCATIONS:
Overall Officials: Terence C Burns, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Riviere-Cazaux C, Rajani K, Rahman M, Oh J, Brown DA, White JF, Himes BT, Jusue-Torres I, Rodriguez M, Warrington AE, Kizilbash SH, Elmquist WF, Burns TC. Methodological and analytical considerations for intra-operative microdialysis. Fluids Barriers CNS. 2023 Dec 19;20(1):94. doi: 10.1186/s12987-023-00497-2. PMID 38115038
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials